CLINICAL TRIAL: NCT03686293
Title: A Personal Microbiome-dependent Glucose Response in Healthy Young Volunteers: a Meal Test Study
Brief Title: A Personal Microbiome-dependent Glucose Response in Healthy Young Volunteers
Acronym: MIGLUCOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M233
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Blood Glucose, High
Keywords: Glucose tolerance; Gut microbiota; Microbial richness; Gastric emptying; Metabolomics

STUDY DESIGN:
Intervention Model Description: Acute meal test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paracetamol and breakfast (Experimental): One tablet of paracetamol (500 mg) and a standardized breakfast will be consumed within 15 minutes one morning upon 10 hours of fasting
  Interventions: Other: Standardized breakfast

INTERVENTIONS:
Other: Standardized breakfast — One tablet of paracetamol (500 mg) and a glass of water (150 mL) is consumed followed by a breakfast consisting of white bread, butter, jam, and juice (300 mL) and

SUMMARY:
Individuals eating identical meals present high variability in post-meal blood glucose response making comparisons challenging. This study evaluates in 40 healthy and fasted participants whether the postprandial glucose response upon a standardized breakfast is dependent on gut microbial richness. Gastric emptying rate, intestinal transit time, insulin, appetite hormones and measures of the intestinal microbiome and fermentation will also be analyzed in the context of postprandial glucose metabolism.

DETAILED DESCRIPTION:
Elevated blood glucose levels constitute a major risk factor for pre-diabetic and diabetic patients. Postprandial glucose tests have been used for decades to monitor and compare glucose responses. Yet, individuals eating identical meals present high variability in post-meal blood glucose response making comparisons challenging. A recent landmark study showed that the inter-individual variation of postprandial glucose responses was associated with multiple person-specific factors including faecal microbiome factors. Gut microbial richness has for a long time been considered a hallmark of gut health and stability. Furthermore, microbial richness has been associated with colonic transit time, which together with the gastric emptying rate appear to be major determinants of the initial glycaemic response to carbohydrate-containing meals. Therefore, the aim of the study is to investigate whether postprandial glucose responses are associated with gut microbial richness, as well as secondary measures including gastric emptying rate, intestinal transit time and gut microbial composition and fermentation.

In an acute-meal study, 40 healthy fasted participants will consume a standardized breakfast including one tablet of paracetamol (for estimating gastric emptying rate) and 300 mL of juice.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 27
* Willing to eat lentils, tomatoes, spaghetti, bread, butter, strawberry jam, and drink juice
* Known ability to tolerate paracetamol
* No current use of medication (oral contraceptive pill and mild antidepressants is allowed)
* Did not take antibiotics, diarrhoea inhibitors and laxatives in the 6 previous months
* Willing to collect and deliver a faecal sample on the intervention day
* Willing to eat corn and fill out a self-reported corn-intestinal transit time questionnaire
* Willing to consume a paracetamol tablet (500 mg paracetamol)

Exclusion Criteria:

* Any condition that makes the project responsible researcher to doubt the feasibility of the volunteer's participation
* Pregnant or lactating women
* Suffering from irritable bowel disease (IBS), small intestine bacterial overgrowth (SIBO) or inflammatory bowel disease (IBD)
* Current chronic or infectious disease
* Current diagnosis of diabetes
* Blood donations within 3 months before participating in the current trial or participation in other scientific experiments
* Frequent intake of painkillers (paracetamol)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Postprandial plasma glucose at 60 min as a function of gut microbial richness | 60 min
  We test whether there is an inverse association between baseline fecal gut microbial richness and postprandial plasma glucose at 60 min after a standardised meal including 0.5 g paracetamol

SECONDARY OUTCOMES:
Fasting (baseline) plasma glucose as a function of gut microbial diversity/richness | 0 min
  We test whether there is an inverse association between fasting plasma glucose and baseline fecal gut microbial richness (cross-sectionally)
Maximum plasma glucose concentration as a function of gut microbial diversity/richness | 0, 15, 30, 60, 90 and 120 min
  We test associations between gut microbial diversity/richness and maximum postprandial plasma glucose concentration [Cmax] after a standardised meal including 0.5 g paracetamol.
Postprandial plasma glucose extremes as a function of gut microbial diversity/richness | 0, 15, 30, 60, 90 and 120 min
  We test associations between gut microbial diversity/richness and the difference from the postprandial plasma glucose peak to the glucose level after 60 min or at the postprandial minimum between 30-120 min after a standardised meal including 0.5 g paracetamol.
Time to plasma glucose maximum concentration as a function of gut microbial diversity/richness | 0, 15, 30, 60, 90 and 120 min
  We test associations between gut microbial diversity/richness and the time to the postprandial plasma glucose maximum concentration [Cmax] after a standardised meal including 0.5 g paracetamol
Postprandial plasma glucose AUC as a function of gut microbial richness/diversity | 0, 15, 30, 60, 90 and 120 min
  We test associations between gut microbial diversity/richness and AUC 0-120 min for plasma glucose after a standardised meal including 0.5 g paracetamol
Postprandial glucose 0-60 min as a function of gastric emptying | 0, 15, 30, 60 min
  We test associations between gastric emptying measured as AUC 0-60 min of postprandial paracetamol concentration profiles in blood and postprandial plasma glucose at 60 min during a standardised meal including 0.5 g paracetamol
Gastric emptying and postprandial glucose 0-120 min | 0, 15, 30, 60, 90 and 120 min
  We test associations between gastric emptying measured as AUC 0-120 min of postprandial paracetamol concentration profiles in blood and postprandial plasma glucose AUC 0-120 min during a standardised meal test with intake of 0.5 g paracetamol

OTHER OUTCOMES:
Saliva microbiome | 0 min
  Determination of saliva microbiome composition at baseline
Fecal microbiome | 0 min
  Determination of fecal microbiome composition at baseline
Urine metabolome | 0, 0-150 min
  Urine metabolome as determined by untargeted metabolic profiling by LC-QTOF of all urine samples collected before the meal and postprandially from 0-150 min
Fecal metabolome | 0 min
  Fecal metabolome as determined by untargeted metabolic profiling by LC-QTOF of ethanolic extracs from all baseline fecal samples collected before the intervention
Plasma metabolome | 0, 15, 30, 60, 90 and 120 min
  Plasma metabolome as determined by untargeted metabolic profiling by LC-QTOF of ethanolic extracs from all fasting and postprandial plasma samples
Glucose metabolism | 0, 15, 30, 60, 90 and 120 min
  Plasma glucose measured in fasting and postprandial plasma samples
Plasma Insulin | 0, 15, 30, 60, 90 and 120 min
  Plasma insulin measured in fasting and postprandial plasma samples
Plasma short-chain fatty acids | 0, 15, 30, 60, 90 and 120 min
  Plasma short-chain fatty acids measured in fasting and postprandial plasma samples
Lipid metabolism | 0, 15, 30, 60, 90 and 120 min
  Bile acids in blood (fasting and postprandially) and in feces (baseline)
Glucagon like peptide 1 (GLP-1) | 0, 15, 30, 60, 90 and 120 min
  Plasma glucagon like peptide 1 (GLP-1) measured in fasting and postprandial plasma samples
Peptide tyrosine tyrosine (PYY) | 0, 15, 30, 60, 90 and 120 min
  PYY measured in fasting and postprandial plasma samples
Ghrelin | 0, 15, 30, 60, 90 and 120 min
  Ghrelin measured in fasting and postprandial plasma samples
Gastric inhibitory polypeptide (GIP) | 0, 15, 30, 60, 90 and 120 min
  GIP measured in fasting and postprandial plasma samples
Cholecystokinin (CCK) | 0, 15, 30, 60, 90 and 120 min
  CCK measured in fasting and postprandial plasma samples
Gastric emptying | 0, 15, 30, 60, 90 and 120 min
  Gastric emptying measured as postprandial paracetamol concentration profiles in blood
Postprandial breath exhalation | 0, 60, 150 min
  Fasting and postprandial breath hydrogen/methane exhalation
Feces short-chain fatty acids | 0 min
  Feces short-chain fatty acids measured in all fecal samples collected at baseline
Feces pH | 0 min
  Feces pH measured in all fecal samples collected at baseline
Feces energy | 0 min
  Feces energy measured in all fecal samples collected at baseline by bomb calorimetry
Stool consistency | 0 min
  Consistency of stool sample collected at baseline assessed by the Bristol stool scale
Intestinal transit time | Before intervention
  Participants are instructed to observe the time it takes corn to travel through their gastrointestinal system five days prior to the intervention
Defecation patterns | Before intervention
  Average number of poops per day and average stool consistency as assessed by Bristol stool scale
Gastrointestinal symptoms | Before intervention
  Gastrointestinal symptoms measured on a 10 cm visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Dragsted, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg, Denmark